CLINICAL TRIAL: NCT05418166
Title: Impact of Evolocumab on the Antiplatelet Effects of Ticagrelor and Aspirin in Patients With Acute Coronary Syndrome
Acronym: EvoACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yongtai Gong
Record Dates: First submitted 2022-06-05; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Evolocumab; Antiplatelet; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — evolocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — about 4ml plasma in -80℃ refrigerator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- pro-Evo: Patients regularly take Ticagrelor and Aspirin for five days.Platelet activity was test before inject Evolocumab.
- 24h-Evo: Patients regularly take Ticagrelor and Aspirin for five days, then inject Evolocumab 140mg. Platelet activity was test 24h after inject.
  Interventions: Drug: Evolocumab
- 1w-Evo: Patients regularly take Ticagrelor and Aspirin for five days, then inject Evolocumab 140mg. Platelet activity was test 1 week after inject.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — evolocumab 140mg subcutaneous injection after regular take Ticagrelor and Aspirin for 5 days.
  Groups: 1w-Evo; 24h-Evo

SUMMARY:
The aim of the present study is to investigate the effects of evolocumab in addition to statin therapy on platelet reactivity in patients with acute coronary syndrome (ACS) while on Ticagrelor and Aspirin treatment.

DETAILED DESCRIPTION:
Ticagrelor is a commercially available antiplatelet adenosine diphosphate (ADP) antagonists. They exert their antiplatelet effects by binding to P2Y12 receptors on the platelet surface. Ticagrelor is used in combination with aspirin to prevent and treat thrombosis in patients with acute coronary syndrome, particularly after stent implantation.

Aspirin has an established role in the treatment of ACS and secondary prevention of ischaemic heart disease. Aspirin inhibits cyclo-oxygenase (COX) enzymes by irreversible acetylation to block platelet aggregation.

Evolocumab is a monoclonal antibody targeting proprotein convertase subtilisin/kexin type 9 (PCSK9). The use of evolocumab significantly reduced the incidence of cardiovascular events compared to statins alone. Whether the reduction in cardiovascular events is due to LDL reduction or other mechanisms is currently unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were diagnosed as acute coronary disease
2. On therapy with Ticagrelor(90mg bid) and Aspirin(100mg qd), for at least 5 days.
3. Fasting LDL-cholesterol ≥70 mg/dL or a non-high-density lipoprotein cholesterol (HDL-C) of ≥100 mg/dL after ≥4 weeks of optimized stable lipid-lowering therapy with maximally tolerated dose of statin.
4. Have not used Evolocumab in 30 days.

Exclusion Criteria:

1. On treatment with any oral anticoagulant.
2. On treatment with any antiplatelet agent other than Aspirin and Ticagrelor in the past 5 days.
3. Creatinine clearance <30 mL/minute.
4. Known severe hepatic impairment.
5. History of a serious hypersensitivity reaction to evolocumab
6. Hemodynamic instability
7. Pregnant and breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the first affiliated hospital of Harbin Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Platelet Reactivity Defined by VerifyNow PU in Patients diagnosed ACS | 1 week
  The primary end point of our study is the comparison of P2Y12 reaction units (PU) measured by VerifyNow in patients before use evolocumab and 24hours after injected and 1week after injected. PU is well-established measures of platelet reactivity and aggregation in response to antiplatelet medications. The higher is the PU the lower is the effect of the antiplatelet medication. Validity is defined as PU<208.
Platelet Reactivity Defined by VerifyNow AU in Patients diagnosed ACS | 1 week
  The second end point of our study is the comparison of COX-1 reaction units(AU) measured by VerifyNow in patients before use evolocumab and 24hours after injected and 1week after injected. AU is well-established measures of platelet reactivity and aggregation in response to antiplatelet medications. The higher is the AU the lower is the effect of the antiplatelet medication. Validity is defined as AU<550.

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Harbin Medical University, Harbin, Heilongjiang, China